CLINICAL TRIAL: NCT03548688
Title: Investigation and Detection of Urological Neoplasia in Patients Referred With Suspected Urinary Tract Cancer: A Multicentre Analysis
Brief Title: Investigation and Detection of Urological Neoplasia in Patients Referred With Suspected Urinary Tract Cancer:
Acronym: IDENTIFY
Status: Completed | Type: Observational
Sponsor: British Urology Researchers in Surgical Training (Other)
Collaborators: The Urology Foundation (Unknown); Action Bladder Cancer UK (Other); Test Evaluation Research Group Birmingham University (Unknown)
Responsible Party: Sponsor
Other Study IDs: IDENTIFY; ABC UK 2017/18 (Other Grant/Funding Number: Action Bladder Cancer UK); TUF Grant 2017 (Other Grant/Funding Number: The Urology Foundation)
Record Dates: First submitted 2018-04-28; First posted 2018-06-07 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Urothelial Carcinoma
Keywords: Bladder Cancer; Haematuria; Collaborative study
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bladder cancer is common in the UK and can kill. A common sign of bladder cancer is blood in the urine (haematuria).

GPs will refer to a specialist (Urologist) for further investigation of haematuria if they suspect cancer.

Hospitals often have a 'blanket' approach for investigating patients with haematuria. IDENTIFY will collect data on patients having these tests across the UK and internationally, looking at any trends with an aim to create a personalised diagnostic approach for each patient. The data will give patients the ability to make informed decisions, as well as reducing unnecessary and potentially harmful tests.

DETAILED DESCRIPTION:
IDENTIFY aims to be the largest contemporary study providing data on the utility of the current diagnostic pathway for bladder and upper urinary tract cancer in patients presenting with haematuria.

It also aims to provide a contemporary evaluation of current urological practices and assessment of the prevalence of urinary tract cancers (bladder cancer, upper tract cancer, renal cancer) in patients with haematuria. This will allow us to recommend changes in cancer diagnosis pathways that may reduce the number of invasive procedures, reduce waste of resources and optimize use of the most appropriate tests. This will mean resources are spent effectively, allowing for early diagnosis and faster treatment pathways.

An evaluation of the patient factors that predict urinary tract cancer, particularly high-risk disease, may allow clinicians to better recognise groups of patients that will benefit from invasive investigations and are more likely to benefit from prompt diagnosis and treatment. Upper tract urinary cancer is quite rare and difficult to diagnose. It requires a large patient cohort such as the IDENTIFY study in order to recognise associations with the diagnosis of this disease and optimize the way we diagnose it.

Shared-decision making is extremely important in patients presenting with haematuria and the outcomes of IDENTIFY will allow a more personalized approach to the diagnosis of urinary tract cancer. For example, rather than a blanket approach in which all patients undergo flexible cystoscopy and one or more imaging tests, we will generate data that could offer patients information on the likelihood of a flexible cystoscopy or other test finding cancer for them, given their personal characteristics.

IDENTIFY results are also hoped to help inform national and international guidelines on referral for haematuria.

ELIGIBILITY:
Inclusion Criteria:

* Any patient referred with haematuria (visible and non-visible) undergoing cystoscopy
* Any patient referred without haematuria undergoing cystoscopy for the purpose of ruling out urothelial cancer suspected due to other symptoms (e.g. lower urinary tract symptoms, recurrent urinary tract symptoms, dysuria)

Exclusion Criteria:

* Patients with a previous or known diagnosis of primary upper or lower urinary tract urothelial cancers (renal, ureteric, bladder, prostate, urethral and penile cancers)
* Patients with suspected recurrence of upper or lower urinary tract primary urothelial cancer (renal, ureteric, bladder, prostate, urethra and penile cancers)
* Patients undergoing flexible cystoscopy for a reason unrelated to ruling out urinary tract urothelial cancer

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to secondary care for further investigation of suspected urinary tract cancer
Sampling Method: Non-Probability Sample
Enrollment: 11059 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence | 12 months
  Determine the prevalence of urological cancers in patients presenting to secondary care with suspected urinary tract cancer

SECONDARY OUTCOMES:
Specific prevalence | 12 months
  Determine the difference in prevalence of urological cancer in those undergoing flexible cystoscopy with visible haematuria, non-visible haematuria and without haematuria
Diagnostic strategies | 12 months
  Describe the current practices in urothelial cancer diagnosis across a range of different healthcare settings in secondary care (district general vs university teaching hospital) with regards to percentage of ultrasound, CT and other imaging modality used for visible and non visible haematuria.
Diagnostic performance of imaging | 12 months
  Determine the diagnostic performance of US, CT, urine cytology and flexible cystoscopy in patients presenting with haematuria in the diagnosis of bladder cancer, using sensitivity, specificity, positive and negative predictive value.
Associated factors | 12 months
  Perform a multivariable analysis to determine factors associated with the diagnosis of bladder cancer and upper urinary tract cancer in patients presenting with haematuria

CONTACTS AND LOCATIONS:
Locations (1):
- BURST, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Country specific data to be given to each country